CLINICAL TRIAL: NCT00335348
Title: Bortezomib and Dexamethasone as Treatment and Maintenance for Multiple Myeloma Relapse An Australian Myeloma Forum Multi-Centre Phase II Trial
Brief Title: Bortezomib and Dexamethasone as Treatment and Maintenance for Multiple Myeloma Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05/69; ACTRN (pending)
Record Dates: First submitted 2006-06-07; First posted 2006-06-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2011-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapse; Bortezomib; Dexamethasone; Maintenance
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bortezomib; Dexamethasone

ARMS (1):
- Bortezomib and Dexamethasone (Experimental)
  Interventions: Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Induction- 1.3mg/m2 IV days 1,4,8,11 every 3 weeks up to 8 cycles Consolidation- 1.3mg/m2 IV days 1,8,15,22 every 5 weeks up to 3 cycles Maintenance- 1.3mg/m2 IV days 1,15 every 4 weeks
Drug: Dexamethasone — Induction- 20mg orally days 1,2,4,5,8,9,11,12 every 3 weeks up to 8 cycles Consolidation- 20mg orally days 1,2,8,9,15,16,22,23 every 5 weeks up to 3 cycles Maintenance- 20mg orally days 1,2,15,16 every 4 weeks

SUMMARY:
This study has two main aims. The first is to assess whether Dexamethasone can increase the number of patients with who respond to Velcade.

The second aim of this study is to see whether treating patients with relapsed multiple myeloma with Velcade and Dexamethasone for a longer period of time extends the time that the myeloma is under control.

DETAILED DESCRIPTION:
Velcade is a new drug, which is being developed for the treatment of patients with a variety of cancers. In studies to date, it has been shown to be useful in the treatment of patients with advanced multiple myeloma whose myeloma has progressed after standard drug treatment. Approximately one third of them have had a response to treatment, which has lasted for approximately 12 months. It has been associated with improvement in symptoms from the disease including improvements in blood counts, fewer blood transfusions and in a lessening of bone pain. There is some evidence that more patients respond to Velcade when it is given together with a steroid drug, Dexamethasone, which is commonly used in the treatment of Myeloma, and you may have received in the past. Only a small number of patients have been treated with Velcade and Dexamethasone from the beginning of therapy. However, many more have had Dexamethasone added later if they have failed to respond to Velcade on its own.

Velcade is approved in the USA and Europe by the Food and Drug Administration (FDA) for the treatment of patients with myeloma. However, Velcade is not approved in Australia and therefore its use in this study is considered experimental.

This study has two main aims. The first is to assess whether Dexamethasone can increase the number of patients who respond to Velcade in the controlled setting of a clinical trial. This study is specifically designed for patients who have received at least one kind of standard treatment in the past and are now in need of further therapy because their disease has relapsed. The second aim of this study is to see whether treating patients with Velcade and Dexamethasone for a longer period of time extends the time that the myeloma is under control. This is known as maintenance treatment.

Approximately 100 patients will participate around Australia.

ELIGIBILITY:
Inclusion Criteria:

* Patient was previously diagnosed with multiple myeloma based on standard criteria and currently requires second or *third line therapy because of PD, defined as a 25% increase in M-protein, or development of new or worsening of existing lytic bone lesions or soft tissue plasmacytomas, or hypercalcemia (serum calcium >11.5 mg/dL), or relapse from CR.*Patients will only be eligible for bortezomib as 3rd line therapy if they have received dexamethasone alone, thalidomide alone (or with corticosteroids) or revlimid alone (or with corticosteroids) as one of the 2 prior therapies.
* Patient is of a legally consenting age, as defined by local regulations.
* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Female patient is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male patient agrees to use an acceptable method for contraception for the duration of the study.
* Patient has measurable disease
* Patient has a Karnofsky performance status ≥60%.
* Patient has a life-expectancy >3 months.

Exclusion Criteria:

* Primary Dexamethasone resistance
* Prior therapy with Bortezomib
* Prior severe allergic reactions to Bortezomib (Velcade), Boron or Mannitol
* Neuropathy > Grade 2 with pain by NCI-CTCAE criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate, defined as the best response on treatment assessed using the EBMT criteria | 2 years

SECONDARY OUTCOMES:
Time To Progression, defined as the time from commencement of treatment to the date of first evidence of progressive disease. | 2 years
Overall survival, defined as the time from commencement of treatment to the date of death from any cause. | 2years

CONTACTS AND LOCATIONS:
Overall Officials: Miles Prince, MD, Principal Investigator — Peter MacCallum Cancer Centre, Melbourne, Australia.; Simon Harrison, MB, BS., PhD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Harrison SJ, Quach H, Link E, Feng H, Dean J, Copeman M, Van De Velde H, Schwarer A, Baker B, Spencer A, Catalano J, Campbell P, Augustson B, Romeril K, Prince HM. The addition of dexamethasone to bortezomib for patients with relapsed multiple myeloma improves outcome but ongoing maintenance therapy has minimal benefit. Am J Hematol. 2015 May;90(5):E86-91. doi: 10.1002/ajh.23967. Epub 2015 Feb 27. PMID 25651830